CLINICAL TRIAL: NCT04499157
Title: Effect of MEMOPTIC on Visual Field of Patients Followed for a Chronic Open-angle Glaucoma
Acronym: MEMO-GCAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2019_843_0061
Record Dates: First submitted 2020-07-29; First posted 2020-08-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Open-angle Glaucoma; Visual Field
Keywords: Citicoline; Gingko biloba; magnesium; Open-angle Glaucoma; visual field; MEMOPTIC
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEMOPTIC added to the usual treatment of glaucoma (Experimental): MEMOPTIC added to the usual treatment of glaucoma
  Interventions: Drug: MEMOPTIC
- usual treatment of glaucoma (Active Comparator): usual treatment of glaucoma
  Interventions: Drug: usual treatment of glaucoma

INTERVENTIONS:
Drug: MEMOPTIC — Patients will receive their usual treatment of glaucoma adding 1 tablet of MEMOPTIC per day during 2 years of following
  Arms: MEMOPTIC added to the usual treatment of glaucoma
Drug: usual treatment of glaucoma — Patients will receive only their usual treatment of glaucoma.
  Arms: usual treatment of glaucoma

SUMMARY:
Open-angle glaucoma is a degeneration of the optic nerve, highlighted by campimetric alterations, and wose only current therapeutic target is the lowering of the intra-ocular pressure (using eye drops, surgery or laser). MEMOPTIC is a tablet combining citicoline, magnesium and Gingko biloba, which have a neuroprotective effect already used in neurodegenerative diseases such as Alzheimer's disease for example. Citicoline has also shown several promising results in ophthalmological diseases (glaucoma, amblyopia or more recently in ischemic optic neuropathies). The citicoline used in eye drops (NEURODROP) has already shown results on the preservation of the vision of glaucomatous patients.

The purpose of this project is to determine if MEMOPTIC can have an effect, in addition to the conventional treatments, in the preservation of vision of patients treated for an open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GCAO defined by OCT RNFL alterations and visual fields defects
* age between 20 and 80 years old
* Well controled intra-ocular pressure under treatment (PIO<21mmHg or decreased by 20% compared to initial the PIO)

Exclusion Criteria:

* retinal or macular disease
* diagnosis of cataract or surgery of cataract during the follow-up
* allergy to citicolin
* ocular hypertonia due to a secondary cause (like corticosteroids)
* history of anterior, intermediate or posterior uveitis
* general treatment affecting PIO (beta blockers, corticosteroids)
* pregnancy or breastfeeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Variation of visual field of open angle-glaucoma patients with MEMOPTIC treatment | from day 0 to 2 years
  Variation of visual field of open angle-glaucoma patients with MEMOPTIC treatment versus visual field of open angle-glaucoma patients without MEMOPTIC treatment. Visual field is measure with METROVISION Visual Field 24-2, a full field projection perimeter entirely compatible with the Goldmann standard and modern perimetry standard. It allows high resolution static perimetry as well as kinetic perimetry with automated and manual modes. Automated static perimetry is one of the methods used to screen and follow up patients who have glaucoma. It consists of approximately 100 quantitative threshold measures that permit evaluation of retinal sensitivity. Each measure is standardized in a population free of ocular disease, and two simple statistics are calculated: mean deviation (MD) and pattern standard deviation (PSD). These indices are widely used in glaucoma clinical trials and patient follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Iscar, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No